CLINICAL TRIAL: NCT02978638
Title: Restoration of Bladder and Bowel Function Using Electrical Stimulation and Block After Spinal Cord Injury
Brief Title: Electrical Stimulation for Continence After Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Stanford University (Other); Case Western Reserve University (Other); Santa Clara Valley Medical Center (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, Graham Creasey, Professor, Palo Alto Veterans Institute for Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE0004AGG; W81XWH-14-2-0132 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury; Neurogenic Bladder; Incontinence
Keywords: Spinal cord injury; Bladder capacity; Electrical stimulation; Continence; Urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Finetech Vocare Bladder System (Other): This is a pilot study of the Finetech Vocare Bladder System to improve continence and voiding in human subjects with chronic spinal cord injury. Each subject will act as their own control, comparing function with the Finetech Vocare Bladder System in use and not in use.
  Interventions: Device: Finetech Vocare Bladder System

INTERVENTIONS:
Device: Finetech Vocare Bladder System — Participants will be implanted with the existing FDA-approved Finetech Vocare Bladder System stimulator and electrodes.

SUMMARY:
This study aims to improve continence and voiding of patients with spinal cord injury using electrical stimulation.

The Finetech Vocare Bladder System is an implantable sacral nerve stimulator for improving bladder and bowel function in patients with spinal cord injury (SCI). It has been commercially available in Britain and other countries since 1982, and has been used in thousands of patients with SCI to improve bladder, bowel and sexual function. It received FDA approval in 1998 under Humanitarian Device Exemption H980005 and H980008 for providing urination on demand and to aid in bowel evacuation.

Electrical stimulation to produce bladder contraction and improve bladder voiding after spinal cord injury has usually been combined with cutting of sensory nerves to reduce reflex contraction of the bladder, which improves continence. However, cutting these nerves has undesirable side effects. This study will not cut any sensory nerve. This study is testing the use of the stimulator for inhibiting bladder contraction by stimulating sensory nerves to improve continence after spinal cord injury, and for blocking sphincter contraction to improve voiding.

DETAILED DESCRIPTION:
Human subjects will be recruited from people with clinically complete spinal cord injury.

Subjects who meet the selection criteria described below will be screened to identify those whose reflex bladder contractions are inhibited by neuromodulation using low levels of electrical stimulation via electrodes on the skin over the dorsal genital nerve. Serial filling cystometries will be performed in the clinical urodynamic laboratories at the study sites. Bladder capacity and compliance will be recorded for each cytometrogram. Subjects whose reflex bladder contractions are significantly inhibited by this neuromodulation will be offered enrollment in the trial. Subjects whose reflex bladder contractions are not significantly inhibited by this neuromodulation, or who do not wish to participate in the study, will be able to continue with their usual form of bladder management.

After screening, selected subjects will be offered surgical implantation of a Vocare Bladder System in the FDA-approved manner, but without posterior rhizotomy. Because posterior rhizotomy is not performed, the afferent axons in the sacral nerves are intact and can be stimulated after surgery via the electrodes connected to the implanted stimulator.

The Vocare Bladder System will be implanted in the FDA-approved manner but without posterior rhizotomy.

After implantation, subjects will be evaluated in the urodynamic laboratory. Stimulation will applied to S34 sacral nerves bilaterally, and the effects on bladder capacity and continence and voiding will be measured.

Continence of urine will be documented by bladder diaries. These diaries will be completed initially as an inpatient in the SCI Service and then at home while applying neuromodulation via the implant.

It is expected that sacral neuromodulation by this method will be associated with a significant increase in bladder capacity and continence.

It is possible that this neuromodulation will not be associated with an increase in bladder capacity or continence. If so, subjects will still be able to use conventional methods of managing continence and should have no loss of function.

Participants whose bladder capacity and continence are improved by neuromodulation using the implanted stimulator will be offered the opportunity to continue to use the stimulator for the duration of the study and will be reviewed at three-month intervals. At the end of the study they will be reviewed again with their usual clinician and if there are no contra-indications to continued use of the stimulator will be offered the opportunity to continue its use under continued clinical follow-up from their usual clinician.

Participants whose bladder capacity and continence are not improved by neuromodulation using the implanted stimulator, or who do not wish to continue using the implanted stimulator, will be reviewed with their usual clinician and offered the bladder management they were using prior to the study. The implanted stimulator will be switched off, but will not be removed unless the participant wishes it to be removed or the investigators or the participant's usual clinician consider it in the participant's interest to be removed. It is usually simpler and safer for the participant to leave the stimulator implanted but inactive.

All participants will be provided with appropriate documentation regarding safety and electromagnetic compatibility of the device.

The investigation is justified because the potential benefits are greater than the potential risks, as follows:

The potential benefit of the research to the subjects are:

1. Improved bladder capacity
2. Improved continence

The potential benefits of the research to others are:

Evidence that bladder capacity and continence after spinal cord injury can be improved by electrical stimulation without cutting nerves.

The risks to subjects are reasonable in relation to the anticipated benefits to subjects and others because of

1. The high prevalence and severity of clinical complications caused by bladder complications after spinal cord injury
2. The paucity of methods of restoring continence after spinal cord injury that are safe, effective and without undesirable side effects

This study is primarily aimed at demonstrating safety, feasibility and proof of concept. It may also produce statistically and clinically significant evidence of efficacy that can be used to plan future clinical trials.

Significance:

If the technique of reducing reflex bladder contraction by implanted stimulation of the S34 nerve bilaterally is successful, it will open the door to more effective use of neuromodulation for continence after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they meet all of the following criteria:

* Complete spinal cord injury (AIS grade A) of at least 2 years duration with neurological level (ISNCSCI level) below C4
* Impaired bladder emptying due to Detrusor External Sphincter Dyssynergia-DESD (unco-ordinated contraction of bladder and external urethral sphincter) as shown on video-urodynamic testing.
* Impaired continence due to detrusor hyper-reflexia

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Absence of reflex contractions of the bladder as shown on urodynamic testing
* Absence of reflex contractions of the external urethral sphincter as shown on urodynamic testing with EMG
* External sphincterotomy, urethral stricture or previous urethral or sphincter or bladder or prostate surgery
* History of pelvic fracture
* Subjects on anticoagulants or with coagulation disorders
* Immunosuppressed subjects
* Active or recurrent pressure ulcers, particularly in sacral, ischial or trochanteric areas
* Active untreated infection
* Active implanted medical device such as cardiac pacemaker or defibrillator
* Progressive spinal cord injury
* Pregnancy
* Mechanical ventilator dependency
* Any other significant co-morbidity or illness that would preclude their participation or increase the risk to them of participating in the study
* Inability or unwillingness to follow study protocol or give informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-09; Primary Completion 2025-08-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Bladder capacity | Change from baseline bladder capacity at 12-month follow-up visit
  Bladder capacity (ml.) measured during filling cystometry

SECONDARY OUTCOMES:
Frequency of incontinence of urine | Change from baseline frequency of incontinence of urine at 12-month follow-up visit
  Frequency of incontinence determined from diary data collected by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Graham H. Creasey, MD, Principal Investigator — Palo Alto Veterans Institute for Research; Reza Ehsanian, MD PhD, Study Director — University of New Mexico
Locations (4):
- United States (4):
  - Palo Alto Veterans Institute for Research, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California
  - University of New Mexico, Albuquerque, New Mexico
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Creasey GH, Grill JH, Korsten M, U HS, Betz R, Anderson R, Walter J; Implanted Neuroprosthesis Research Group. An implantable neuroprosthesis for restoring bladder and bowel control to patients with spinal cord injuries: a multicenter trial. Arch Phys Med Rehabil. 2001 Nov;82(11):1512-9. doi: 10.1053/apmr.2001.25911. PMID 11689969
- [Background] Kirkham AP, Knight SL, Craggs MD, Casey AT, Shah PJ. Neuromodulation through sacral nerve roots 2 to 4 with a Finetech-Brindley sacral posterior and anterior root stimulator. Spinal Cord. 2002 Jun;40(6):272-81. doi: 10.1038/sj.sc.3101278. PMID 12037708
- [Background] Kutzenberger J, Domurath B, Sauerwein D. Spastic bladder and spinal cord injury: seventeen years of experience with sacral deafferentation and implantation of an anterior root stimulator. Artif Organs. 2005 Mar;29(3):239-41. doi: 10.1111/j.1525-1594.2005.29043.x. PMID 15725225
- [Background] Martens FM, den Hollander PP, Snoek GJ, Koldewijn EL, van Kerrebroeck PE, Heesakkers JP. Quality of life in complete spinal cord injury patients with a Brindley bladder stimulator compared to a matched control group. Neurourol Urodyn. 2011 Apr;30(4):551-5. doi: 10.1002/nau.21012. Epub 2011 Feb 15. PMID 21328472
- [Background] Martens FM, Heesakkers JP. Clinical results of a brindley procedure: sacral anterior root stimulation in combination with a rhizotomy of the dorsal roots. Adv Urol. 2011;2011:709708. doi: 10.1155/2011/709708. Epub 2011 Jun 22. PMID 21738530
- [Background] Rasmussen MM, Kutzenberger J, Krogh K, Zepke F, Bodin C, Domurath B, Christensen P. Sacral anterior root stimulation improves bowel function in subjects with spinal cord injury. Spinal Cord. 2015 Apr;53(4):297-301. doi: 10.1038/sc.2015.2. Epub 2015 Jan 20. PMID 25600307
- [Background] Schurch B, Rodic B, Jeanmonod D. Posterior sacral rhizotomy and intradural anterior sacral root stimulation for treatment of the spastic bladder in spinal cord injured patients. J Urol. 1997 Feb;157(2):610-4. PMID 8996369
- [Background] van der Aa HE, Alleman E, Nene A, Snoek G. Sacral anterior root stimulation for bladder control: clinical results. Arch Physiol Biochem. 1999 Jul;107(3):248-56. doi: 10.1076/apab.107.3.248.4330. PMID 10650355
- [Background] Van Kerrebroeck PE, Koldewijn EL, Rosier PF, Wijkstra H, Debruyne FM. Results of the treatment of neurogenic bladder dysfunction in spinal cord injury by sacral posterior root rhizotomy and anterior sacral root stimulation. J Urol. 1996 Apr;155(4):1378-81. doi: 10.1097/00005392-199604000-00069. PMID 8632580
- [Background] Vastenholt JM, Snoek GJ, Buschman HP, van der Aa HE, Alleman ER, Ijzerman MJ. A 7-year follow-up of sacral anterior root stimulation for bladder control in patients with a spinal cord injury: quality of life and users' experiences. Spinal Cord. 2003 Jul;41(7):397-402. doi: 10.1038/sj.sc.3101465. PMID 12815371
- [Background] Wielink G, Essink-Bot ML, van Kerrebroeck PE, Rutten FF. Sacral rhizotomies and electrical bladder stimulation in spinal cord injury. 2. Cost-effectiveness and quality of life analysis. Dutch Study Group on Sacral Anterior Root Stimulation. Eur Urol. 1997;31(4):441-6. doi: 10.1159/000474504. PMID 9187905
- [Background] Kirkham AP, Shah NC, Knight SL, Shah PJ, Craggs MD. The acute effects of continuous and conditional neuromodulation on the bladder in spinal cord injury. Spinal Cord. 2001 Aug;39(8):420-8. doi: 10.1038/sj.sc.3101177. PMID 11512072
- [Derived] Ehsanian R, Creasey G, Elliott CS, Abu-Eid CA, Ali A, Prutton M, Singh H. Implantation of Sacral Nerve Stimulator Without Rhizotomy for Neurogenic Bladder in Patient With Spinal Cord Injury: 2-Dimensional Operative Video. Oper Neurosurg. 2020 Sep 1;19(3):E299. doi: 10.1093/ons/opz429. PMID 31980830